CLINICAL TRIAL: NCT02363998
Title: A Phase 3, Open-Label, Safety Study of Lofexidine
Brief Title: Open-Label, Safety Study of Lofexidine
Acronym: NU LEAF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: USWM, LLC (dba US WorldMeds) (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USWM-LX1-3003-2; 1U01DA033276-01A1 (NIH)
Record Dates: First submitted 2015-02-09; First posted 2015-02-16 (Estimated); Results first posted 2021-04-26 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Opioid Withdrawal
Keywords: detoxification; agonist taper; methadone step down; buprenorphine step down; opioid withdrawal syndrome
MeSH Terms: interventions — lofexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label Lofexidine (Other): During this open-label study, subjects will be given the option to receive lofexidine tablets for 7 days and up to 14 days if requested.
  Interventions: Drug: Lofexidine

INTERVENTIONS:
Drug: Lofexidine — All enrolled subjects will take lofexidine orally for 7 days, starting on Day 1 at a dose of 3.2 mg per day (0.8 mg QID), with lowering of the dose allowed to 2.4 mg daily (0.6 mg QID) if required for tolerability based on the subject's individual treatment goal and response per clinical judgment of the Principal Investigator.
  Other Names: Lofexidine hydrochloride (HCL)

SUMMARY:
The purpose of this Phase 3 open-label treatment study is to evaluate the safety and effectiveness of lofexidine at a clinically relevant dose to alleviate symptoms of acute withdrawal from any opioid, including methadone and buprenorphine. This study will take place in a variety of clinical scenarios, both in-clinic and outpatient settings.

DETAILED DESCRIPTION:
Eligible subjects (person seeking treatment for partial or total opioid withdrawal) enrolled in this study are required to take lofexidine for a minimum of 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female at least 18 years of age
* Must be able to verbalize understanding of the consent form, able to provide written informed consent, and verbalize willingness to complete study procedures
* Must have current dependence, according to the Mini International Neuropsychiatric Interview (M.I.N.I.), on any opioid (including methadone and buprenorphine maintenance treatment)
* Must be seeking treatment for partial or total withdrawal from current opioid and expected, as determined by the Principal Investigator, to benefit from lofexidine treatment for at least 7 days at clinically relevant doses. This can include a variety of clinical situations where opioid withdrawal illness is likely to occur including abrupt and total withdrawal (including from methadone and buprenorphine), agonist-assisted total withdrawal, dose reduction of maintenance treatment (e.g., methadone, buprenorphine) and transition from an opioid agonist to naltrexone or buprenorphine maintenance
* Must have Urine toxicology screen result of positive for opioid(s) relevant to the subject's withdrawal treatment goal
* If female and of childbearing potential, subject must agree to use of one of the following methods of birth control including oral contraceptives, patch, barrier (diaphragm, sponge or condom) plus spermicidal preparations, intrauterine contraceptive system, levonorgestrel implant, medroxyprogesterone acetate contraceptive injection, complete abstinence from sexual intercourse, hormonal vaginal contraceptive ring or surgical sterilization or partner sterile (with documented proof)

Exclusion Criteria:

* Female subject who is pregnant or lactating
* History of very serious medical illness not under control including, but not limited to, active self-reported acquired immune deficiency syndrome (AIDS) or self-reported human immunodeficiency virus (HIV) positive status and taking retroviral medications currently or within the past 4 weeks and/or having an unstable psychiatric condition. These conditions will be determined at Screening by medical history, physical examination, 12 lead electrocardiogram (duplicate), clinical laboratory tests for infectious diseases, and a tuberculin test
* Current dependence (based on the M.I.N.I.) on any psychoactive substance (excluding caffeine, nicotine, and the subject's current opioid-dependence agent, which can include methadone and buprenorphine, for example, in agonist-maintained subjects) that requires detoxification or dose reduction as part of the pre-defined individual subject withdrawal treatment goal
* Have participated in an investigational drug study within the past 30 days
* Have a history of lofexidine exposure in a prior clinical trial or otherwise
* Have an abnormal cardiovascular exam at screening
* Any subject that requires tricyclic antidepressants, which may reduce the efficacy of imidazoline derivatives and/or beta-receptor blockers, to avoid the risk of excessive bradycardia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Gorodetzky, MD, PhD, Study Director — US WorldMeds
Locations (18):
- United States (18):
  - Little Rock, Arkansas
  - Springdale, Arkansas
  - San Diego, California
  - Fort Lauderdale, Florida
  - Hollywood, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Winfield, Illinois
  - Lake Charles, Louisiana
  - Rockville, Maryland
  - Flowood, Mississippi
  - St Louis, Missouri
  - New York, New York
  - Dayton, Ohio
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - North Charleston, South Carolina
  - Orem, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- OL: Lofexidine HCl: Lofexidine: All enrolled subjects will take lofexidine orally, starting on Day 1 at a dose of 3.2 mg per day (0.8 mg QID), with lowering of the dose allowed to 2.4 mg daily (0.6 mg QID) if required for tolerability based on the subject's individual treatment goal and response per clinical judgment of the Principal Investigator.
  Subjects are given the option to receive lofexidine tablets for a minimum of 7 days, and up to 14 days if requested.
Period: Overall Study
Arm/Group | OL: Lofexidine HCl
Started | 286
Completed | 168 (A subject was defined as completed if at least one dose was taken on Day 7.)
Not Completed | 118

BASELINE CHARACTERISTICS:
Arm/Group | OL: Lofexidine HCl
Number analyzed (Participants) | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44
  Not Hispanic or Latino | 242
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 62
  White | 218
  More than one race | 0
  Unknown or Not Reported | 5
Height (cm) [Mean (Standard Deviation); unit: cm] | 173.2 (9.99)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 78.4 (17.96)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 26.1 (5.43)

OUTCOME MEASURES:

1. Primary Outcome: Overall Occurrence of Treatment Emergent Adverse Events (TEAEs)
Description: Subjects with at least 1 TEAE occurring on days 1-14.
Time Frame: Days 1-14
Measure: Count of Participants; unit: Participants
Groups:
- OL: Lofexidine HCl: Lofexidine: All enrolled subjects will take lofexidine orally, starting on Day 1 at a dose of 3.2 mg per day (0.8 mg QID), with lowering of the dose allowed to 2.4 mg daily (0.6 mg QID) if required for tolerability based on the subject's individual treatment goal and response per clinical judgment of the Principal Investigator.
Arm/Group | OL: Lofexidine HCl
Number analyzed (Participants) | 286
Participants | 270

2. Primary Outcome: Overall Occurrence of Serious Treatment Emergent Adverse Events (Serious TEAEs)
Time Frame: Days 1-14
Measure: Count of Participants; unit: Participants
Arm/Group | OL: Lofexidine HCl
Number analyzed (Participants) | 286
Participants | 2

3. Primary Outcome: Overall Treatment Emergent Adverse Events (TEAEs) by Severity
Time Frame: Days 1-14
Measure: Count of Participants; unit: Participants
Arm/Group | OL: Lofexidine HCl
Number analyzed (Participants) | 286
Participants
  Mild | 104
  Moderate | 158
  Severe | 8

4. Primary Outcome: Occurrence of Per Protocol Adverse Events of Special Interest (AESI)
Time Frame: Day 1 to Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | OL: Lofexidine HCl
Number analyzed (Participants) | 286
Participants
  Orthostatic hypotension | 96
  Orthostatic bradycardia | 0
  Syncope | 1

5. Primary Outcome: Occurrence of Adverse Events (AEs) Not Related to Opioid Withdrawal
Time Frame: Day 1 to Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | OL: Lofexidine HCl
Number analyzed (Participants) | 286
Participants
  Opioid Withdrawal Related Adverse Events | 233
  Non-Opioid Withdrawal Related Adverse Events | 208

6. Primary Outcome: Mean Observed and Change From Screening in Seated Systolic Blood Pressure (mmHg): Vital Sign
Description: Baseline vital signs were defined by the assessment value at screening when subjects were not experiencing opioid withdrawal to reduce the potential for variability from the effects of different states of withdrawal that may have been present before dosing on Day 1.
  Overall screening values are captured in the column "Inpatient: Pre 8AM"; these values were recorded at various times for each participant during the screening visit, not necessarily at 8AM.
  Serial vital sign assessments required for inpatient visits on days 1-3, either inpatient or outpatient for days 4-7, and outpatient only for days 8-14.
  Day 14 only required pre-dose vital signs measurement. Day 1 Change, Pre 8AM was prior to the first dose.
Time Frame: Day 1 to Day 14
Population: Participants Analyzed does not match the Participant Flow because some patient data was missing for the visit.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Inpatient: Pre 8AM; Inpatient: 3.5 hr Post 8AM; Inpatient: Pre 1PM; Inpatient: 3.5 hr Post 1PM; Inpatient: Pre 6PM; Inpatient: 3.5 hr Post 6PM; Inpatient: Pre 11PM; Outpatient: Predose; Outpatient: 3.5 hr Postdose: Lofexidine: All enrolled subjects will take lofexidine orally for 7 days, starting on Day 1 at a dose of 3.2 mg per day (0.8 mg QID), with lowering of the dose allowed to 2.4 mg daily (0.6 mg QID) if required for tolerability based on the subject's individual treatment goal and response per clinical judgment of the Principal Investigator.
Arm/Group | Inpatient: Pre 8AM | Inpatient: 3.5 hr Post 8AM | Inpatient: Pre 1PM | Inpatient: 3.5 hr Post 1PM | Inpatient: Pre 6PM | Inpatient: 3.5 hr Post 6PM | Inpatient: Pre 11PM | Outpatient: Predose | Outpatient: 3.5 hr Postdose
Number analyzed (Participants) | 286 | 286 | 286 | 286 | 286 | 286 | 286 | 286 | 286
mmHg
  Screening: number analyzed (Participants) | 286 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Screening | 121.9 (11.85) |  |  |  |  |  |  |  |
  Day 1 Observed: number analyzed (Participants) | 286 | 285 | 283 | 270 | 266 | 259 | 257 | 0 | 0
  Day 1 Observed | 122.2 (13.89) | 109.7 (15.47) | 111.1 (16.07) | 112.6 (15.91) | 114.1 (15.38) | 116.9 (17.94) | 116.7 (16.82) |  |
  Day 1 Change: number analyzed (Participants) | 0 | 285 | 283 | 270 | 266 | 259 | 257 | 0 | 0
  Day 1 Change |  | -12.2 (15.25) | -10.8 (15.21) | -9.4 (16.05) | -8.0 (15.12) | -5.2 (19.16) | -5.3 (17.69) |  |
  Day 2 Observed: number analyzed (Participants) | 251 | 235 | 226 | 218 | 217 | 214 | 213 | 0 | 0
  Day 2 Observed | 116.8 (15.77) | 114.8 (15.82) | 114.5 (14.30) | 115.7 (16.20) | 117.4 (16.55) | 119.7 (18.01) | 117.9 (16.04) |  |
  Day 2 Change: number analyzed (Participants) | 251 | 235 | 226 | 218 | 217 | 214 | 213 | 0 | 0
  Day 2 Change | -5.0 (16.21) | -7.0 (15.65) | -7.3 (15.53) | -6.2 (16.43) | -4.5 (17.10) | -2.1 (18.03) | -3.9 (17.24) |  |
  Day 3 Observed: number analyzed (Participants) | 213 | 208 | 206 | 203 | 203 | 203 | 202 | 0 | 0
  Day 3 Observed | 116.0 (15.66) | 116.1 (15.75) | 114.3 (14.71) | 116.9 (16.21) | 116.9 (15.90) | 118.2 (16.64) | 117.1 (15.70) |  |
  Day 3 Change: number analyzed (Participants) | 213 | 208 | 206 | 203 | 203 | 203 | 202 | 0 | 0
  Day 3 Change | -5.9 (16.38) | -5.8 (16.22) | -7.5 (16.40) | -5.0 (17.30) | -5.0 (16.88) | -3.8 (17.08) | -4.9 (16.17) |  |
  Day 4 Observed: number analyzed (Participants) | 161 | 158 | 149 | 144 | 140 | 137 | 133 | 39 | 37
  Day 4 Observed | 116.2 (15.32) | 113.7 (14.26) | 114.4 (14.85) | 118.6 (14.77) | 118.7 (14.68) | 120.0 (15.24) | 117.7 (13.90) | 117.0 (12.44) | 115.7 (8.60)
  Day 4 Change: number analyzed (Participants) | 168 | 162 | 149 | 144 | 140 | 137 | 133 | 286 | 286
  Day 4 Change | -6.0 (15.47) | -8.1 (14.65) | -7.7 (14.77) | -3.7 (15.31) | -3.0 (15.24) | -1.8 (16.36) | -4.0 (16.10) | -4.7 (14.54) | -5.5 (11.15)
  Day 5 Observed: number analyzed (Participants) | 134 | 134 | 132 | 132 | 131 | 129 | 129 | 50 | 46
  Day 5 Observed | 115.4 (14.76) | 114.8 (15.06) | 115.2 (13.69) | 116.3 (15.72) | 117.1 (14.78) | 117.2 (14.62) | 117.0 (13.48) | 116.7 (12.12) | 118.3 (11.06)
  Day 5 Change: number analyzed (Participants) | 139 | 135 | 132 | 132 | 131 | 129 | 129 | 50 | 46
  Day 5 Change | -6.3 (15.86) | -7.1 (16.87) | -6.6 (15.46) | -5.6 (16.76) | -4.8 (16.64) | -4.8 (15.46) | -4.9 (14.93) | -6.3 (16.02) | -4.7 (14.97)
  Day 6 Observed: number analyzed (Participants) | 127 | 126 | 122 | 122 | 121 | 120 | 119 | 50 | 44
  Day 6 Observed | 115.2 (16.13) | 113.4 (14.81) | 114.0 (14.52) | 116.8 (16.74) | 116.6 (15.03) | 117.5 (16.57) | 118.4 (16.46) | 118.7 (15.19) | 122.0 (15.14)
  Day 6 Change: number analyzed (Participants) | 135 | 128 | 122 | 122 | 121 | 120 | 119 | 50 | 44
  Day 6 Change | -6.5 (15.89) | -8.7 (14.74) | -8.0 (14.88) | -5.1 (16.57) | -5.5 (15.10) | -4.5 (17.13) | -3.5 (15.41) | -3.6 (18.44) | 0.4 (19.39)
  Day 7 Observed: number analyzed (Participants) | 114 | 67 | 29 | 27 | 25 | 25 | 24 | 49 | 27
  Day 7 Observed | 118.0 (16.44) | 116.4 (14.82) | 114.9 (15.45) | 117.9 (11.32) | 117.9 (12.20) | 121.1 (14.84) | 118.5 (12.08) | 120.8 (12.99) | 116.3 (9.96)
  Day 7 Change: number analyzed (Participants) | 136 | 67 | 29 | 27 | 25 | 25 | 24 | 49 | 27
  Day 7 Change | -4.4 (16.50) | -5.4 (14.82) | -5.1 (12.87) | -3.0 (13.44) | -3.0 (11.43) | 0.2 (15.23) | -1.7 (16.30) | 2.6 (16.29) | -5.1 (12.91)
  Day 8 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 38
  Day 8 Observed |  |  |  |  |  |  |  | 118.4 (11.69) | 122.8 (13.15)
  Day 8 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 38
  Day 8 Change |  |  |  |  |  |  |  | -2.8 (14.03) | 2.1 (13.41)
  Day 9 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39 | 36
  Day 9 Observed |  |  |  |  |  |  |  | 124.3 (13.14) | 122.3 (16.51)
  Day 9 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39 | 36
  Day 9 Change |  |  |  |  |  |  |  | 3.6 (14.43) | 1.4 (14.75)
  Day 10 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 36 | 34
  Day 10 Observed |  |  |  |  |  |  |  | 122.2 (14.41) | 124.3 (17.24)
  Day 10 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 36 | 34
  Day 10 Change |  |  |  |  |  |  |  | 1.2 (14.12) | 3.6 (17.67)
  Day 11 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 28
  Day 11 Observed |  |  |  |  |  |  |  | 121.2 (12.54) | 125.1 (14.16)
  Day 11 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 28
  Day 11 Change |  |  |  |  |  |  |  | 0.7 (13.52) | 4.6 (15.39)
  Day 12 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 22
  Day 12 Observed |  |  |  |  |  |  |  | 126.3 (9.75) | 120.4 (12.22)
  Day 12 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 22
  Day 12 Change |  |  |  |  |  |  |  | 4.3 (9.20) | -1.4 (12.10)
  Day 13 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20
  Day 13 Observed |  |  |  |  |  |  |  | 124.8 (12.48) | 123.5 (10.61)
  Day 13 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20
  Day 13 Change |  |  |  |  |  |  |  | 4.0 (13.62) | 3.0 (14.38)
  Day 14 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0
  Day 14 Observed |  |  |  |  |  |  |  | 128.0 (12.62) |
  Day 14 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0
  Day 14 Change |  |  |  |  |  |  |  | 7.6 (10.80) |

7. Primary Outcome: Mean Observed and Change From Screening in Standing Systolic Blood Pressure (mmHg): Vital Sign
Description: as for outcome 6
Time Frame: Day 1 to Day 14
Population: Participant Number Analyzed does not match the Participant Flow because some patient data was not captured for the visit.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Inpatient: Pre 8AM | Inpatient: 3.5 hr Post 8AM | Inpatient: Pre 1PM | Inpatient: 3.5 hr Post 1PM | Inpatient: Pre 6PM | Inpatient: 3.5 hr Post 6PM | Inpatient: Pre 11PM | Outpatient: Predose | Outpatient: 3.5 hr Postdose
Number analyzed (Participants) | 286 | 286 | 286 | 286 | 286 | 286 | 286 | 286 | 286
mmHg
  Day 1 Observed: number analyzed (Participants) | 286 | 280 | 281 | 269 | 265 | 258 | 256 | 0 | 0
  Day 1 Observed | 120.4 (13.94) | 105.7 (16.70) | 107.9 (16.43) | 106.7 (15.66) | 108.2 (16.37) | 108.7 (15.75) | 109.0 (16.93) |  |
  Day 1 Change: number analyzed (Participants) | 0 | 279 | 286 | 268 | 264 | 257 | 255 | 0 | 0
  Day 1 Change |  | -16.8 (16.80) | -14.3 (15.95) | -15.8 (16.48) | -14.7 (15.80) | -13.9 (17.31) | -13.6 (17.74) |  |
  Day 2 Observed: number analyzed (Participants) | 251 | 235 | 226 | 218 | 216 | 212 | 213 | 0 | 0
  Day 2 Observed | 112.4 (15.85) | 108.5 (15.94) | 108.0 (15.06) | 108.6 (16.90) | 109.8 (16.22) | 110.4 (17.70) | 110.7 (16.07) |  |
  Day 2 Change: number analyzed (Participants) | 250 | 234 | 225 | 217 | 215 | 211 | 212 | 0 | 0
  Day 2 Change | -10.0 (16.32) | -14.0 (17.24) | -14.7 (16.29) | -14.1 (17.11) | -13.0 (17.07) | -12.2 (17.69) | -11.9 (16.91) |  |
  Day 3 Observed: number analyzed (Participants) | 213 | 207 | 206 | 203 | 203 | 203 | 201 | 0 | 0
  Day 3 Observed | 111.2 (16.61) | 108.1 (17.15) | 109.1 (15.40) | 107.8 (15.97) | 110.0 (15.99) | 110.8 (15.77) | 110.5 (16.19) |  |
  Day 3 Change: number analyzed (Participants) | 212 | 206 | 205 | 202 | 202 | 202 | 200 | 0 | 0
  Day 3 Change | -11.4 (16.25) | -14.4 (17.22) | -13.5 (15.73) | -14.8 (17.63) | -12.6 (17.16) | -11.9 (16.61) | -12.2 (16.09) |  |
  Day 4 Observed: number analyzed (Participants) | 161 | 158 | 149 | 144 | 140 | 137 | 133 | 39 | 37
  Day 4 Observed | 112.4 (15.93) | 107.9 (16.18) | 110.9 (17.93) | 109.7 (14.74) | 112.4 (15.12) | 111.7 (15.81) | 111.1 (14.79) | 116.6 (15.11) | 113.4 (11.60)
  Day 4 Change: number analyzed (Participants) | 160 | 157 | 148 | 143 | 139 | 136 | 132 | 39 | 37
  Day 4 Change | -10.3 (15.29) | -14.4 (15.07) | -11.9 (16.69) | -13.2 (15.66) | -9.9 (15.25) | -10.8 (16.21) | -11.3 (15.89) | -6.1 (17.61) | -8.8 (13.77)
  Day 5 Observed: number analyzed (Participants) | 134 | 134 | 132 | 132 | 131 | 129 | 129 | 50 | 46
  Day 5 Observed | 111.3 (15.97) | 108.9 (15.41) | 109.2 (14.75) | 109.5 (15.75) | 110.8 (14.72) | 110.2 (16.55) | 111.4 (15.49) | 114.6 (12.29) | 116.1 (10.69)
  Day 5 Change: number analyzed (Participants) | 133 | 133 | 131 | 131 | 130 | 128 | 128 | 50 | 46
  Day 5 Change | -11.1 (15.19) | -13.6 (15.83) | -13.2 (16.10) | -13.0 (17.91) | -11.7 (16.44) | -12.3 (17.23) | -11.0 (16.42) | -8.4 (14.43) | -7.5 (15.02)
  Day 6 Observed: number analyzed (Participants) | 127 | 126 | 122 | 122 | 121 | 120 | 119 | 50 | 44
  Day 6 Observed | 112.2 (16.44) | 108.8 (15.61) | 110.2 (15.25) | 109.1 (16.83) | 110.7 (16.44) | 110.9 (16.91) | 112.7 (16.24) | 116.6 (15.47) | 116.4 (16.05)
  Day 6 Change: number analyzed (Participants) | 126 | 125 | 121 | 121 | 120 | 119 | 118 | 50 | 44
  Day 6 Change | -10.4 (16.12) | -14.0 (17.01) | -12.6 (15.30) | -13.8 (17.45) | -12.3 (16.78) | -12.0 (17.84) | -10.0 (16.10) | -5.8 (17.68) | -5.8 (18.68)
  Day 7 Observed: number analyzed (Participants) | 114 | 67 | 29 | 27 | 25 | 25 | 24 | 49 | 27
  Day 7 Observed | 113.9 (17.10) | 113.9 (14.96) | 110.1 (17.41) | 110.1 (15.32) | 112.7 (13.26) | 114.6 (16.42) | 111.6 (14.00) | 118.0 (13.00) | 116.6 (15.53)
  Day 7 Change: number analyzed (Participants) | 113 | 66 | 28 | 26 | 24 | 24 | 23 | 49 | 27
  Day 7 Change | -8.7 (17.74) | -8.2 (16.40) | -8.8 (16.55) | -9.6 (17.71) | -6.8 (14.10) | -4.6 (17.96) | -7.3 (17.01) | -4.6 (15.53) | -5.8 (19.56)
  Day 8 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 38
  Day 8 Observed |  |  |  |  |  |  |  | 117.8 (11.13) | 117.6 (13.94)
  Day 8 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 38
  Day 8 Change |  |  |  |  |  |  |  | -2.8 (13.53) | -2.5 (18.18)
  Day 9 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39 | 36
  Day 9 Observed |  |  |  |  |  |  |  | 119.4 (10.62) | 119.5 (17.05)
  Day 9 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39 | 36
  Day 9 Change |  |  |  |  |  |  |  | -0.8 (13.27) | -0.9 (21.35)
  Day 10 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 36 | 34
  Day 10 Observed |  |  |  |  |  |  |  | 122.3 (14.78) | 121.9 (18.78)
  Day 10 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 36 | 34
  Day 10 Change |  |  |  |  |  |  |  | 1.6 (15.46) | 1.6 (22.89)
  Day 11 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 28
  Day 11 Observed |  |  |  |  |  |  |  | 123.7 (14.91) | 123.2 (14.43)
  Day 11 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 28
  Day 11 Change |  |  |  |  |  |  |  | 3.0 (16.20) | 1.8 (18.90)
  Day 12 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 22
  Day 12 Observed |  |  |  |  |  |  |  | 124.3 (11.19) | 118.4 (14.06)
  Day 12 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 22
  Day 12 Change |  |  |  |  |  |  |  | 2.0 (12.76) | -4.1 (16.91)
  Day 13 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20
  Day 13 Observed |  |  |  |  |  |  |  | 122.7 (11.77) | 125.1 (12.25)
  Day 13 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20
  Day 13 Change |  |  |  |  |  |  |  | 1.0 (14.58) | 3.5 (16.41)
  Day 14 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0
  Day 14 Observed |  |  |  |  |  |  |  | 128.8 (9.89) |
  Day 14 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0
  Day 14 Change |  |  |  |  |  |  |  | 7.8 (9.92) |

8. Primary Outcome: Mean Observed and Change From Screening in Seated Diastolic Blood Pressure (mmHg): Vital Sign
Description: as for outcome 6
Time Frame: Day 1 to Day 14
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Inpatient: Pre 8AM | Inpatient: 3.5 hr Post 8AM | Inpatient: Pre 1PM | Inpatient: 3.5 hr Post 1PM | Inpatient: Pre 6PM | Inpatient: 3.5 hr Post 6PM | Inpatient: Pre 11PM | Outpatient: Predose | Outpatient: 3.5 hr Postdose
Number analyzed (Participants) | 286 | 286 | 286 | 286 | 286 | 286 | 286 | 286 | 286
mmHg
  Day 1 Observed: number analyzed (Participants) | 286 | 285 | 283 | 270 | 266 | 259 | 257 | 0 | 0
  Day 1 Observed | 78.3 (8.89) | 69.4 (10.95) | 69.3 (10.34) | 70.8 (11.13) | 71.5 (10.76) | 73.5 (12.18) | 72.8 (12.26) |  |
  Day 1 Change: number analyzed (Participants) | 286 | 285 | 283 | 270 | 266 | 259 | 257 | 0 | 0
  Day 1 Change | NA (NA) — Prior to first dose. | -7.8 (10.78) | -7.9 (9.88) | -6.3 (11.49) | -5.7 (10.80) | -3.7 (12.52) | -4.3 (12.55) |  |
  Day 2 Observed: number analyzed (Participants) | 251 | 235 | 226 | 218 | 217 | 214 | 213 | 0 | 0
  Day 2 Observed | 73.8 (10.49) | 72.2 (10.89) | 72.2 (10.20) | 73.4 (11.53) | 73.7 (12.08) | 75.4 (11.67) | 74.0 (11.44) |  |
  Day 2 Change: number analyzed (Participants) | 251 | 235 | 226 | 218 | 217 | 214 | 213 | 0 | 0
  Day 2 Change | -3.3 (10.73) | -4.9 (11.17) | -5.0 (10.61) | -3.8 (11.38) | -3.4 (12.04) | -1.8 (12.19) | -3.3 (12.11) |  |
  Day 3 Observed: number analyzed (Participants) | 213 | 208 | 206 | 203 | 203 | 203 | 202 | 0 | 0
  Day 3 Observed | 73.7 (11.05) | 73.2 (10.59) | 71.4 (10.05) | 73.0 (10.48) | 72.9 (10.64) | 73.2 (11.32) | 73.5 (11.08) |  |
  Day 3 Change: number analyzed (Participants) | 213 | 208 | 206 | 203 | 203 | 203 | 202 | 0 | 0
  Day 3 Change | -3.6 (11.60) | -4.0 (10.97) | -5.8 (10.88) | -4.1 (10.32) | -4.3 (10.56) | -4.0 (11.41) | -3.8 (11.37) |  |
  Day 4 Observed: number analyzed (Participants) | 161 | 158 | 149 | 144 | 140 | 137 | 133 | 39 | 37
  Day 4 Observed | 73.9 (10.55) | 71.4 (10.28) | 70.9 (11.11) | 74.7 (10.39) | 73.7 (10.10) | 74.0 (10.95) | 73.4 (9.78) | 75.0 (8.57) | 71.7 (8.53)
  Day 4 Change: number analyzed (Participants) | 161 | 158 | 149 | 144 | 140 | 137 | 133 | 39 | 37
  Day 4 Change | -3.2 (11.06) | -5.7 (10.75) | -6.4 (10.48) | -2.6 (10.27) | -3.3 (9.74) | -3.1 (11.75) | -3.6 (10.51) | -3.0 (10.65) | -6.1 (10.68)
  Day 5 Observed: number analyzed (Participants) | 134 | 134 | 132 | 132 | 131 | 129 | 129 | 50 | 46
  Day 5 Observed | 73.2 (10.42) | 71.5 (10.25) | 71.7 (10.38) | 72.7 (10.58) | 71.8 (10.14) | 73.1 (9.97) | 72.3 (10.44) | 72.6 (9.99) | 72.8 (10.67)
  Day 5 Change: number analyzed (Participants) | 134 | 134 | 132 | 132 | 131 | 129 | 129 | 50 | 46
  Day 5 Change | -3.8 (11.17) | -5.4 (11.75) | -5.1 (10.59) | -4.2 (10.38) | -5.0 (10.79) | -3.7 (10.77) | -4.7 (10.56) | -5.6 (11.18) | -6.0 (12.01)
  Day 6 Observed: number analyzed (Participants) | 127 | 126 | 122 | 122 | 121 | 120 | 119 | 50 | 44
  Day 6 Observed | 72.2 (10.33) | 69.8 (10.46) | 70.8 (10.81) | 72.2 (10.08) | 72.6 (11.02) | 72.8 (11.35) | 72.0 (11.29) | 74.2 (11.25) | 76.8 (9.99)
  Day 6 Change: number analyzed (Participants) | 127 | 126 | 122 | 122 | 121 | 120 | 119 | 50 | 44
  Day 6 Change | -4.6 (9.87) | -7.0 (10.86) | -6.0 (11.42) | -4.6 (10.46) | -4.3 (10.77) | -4.0 (11.05) | -4.9 (11.51) | -3.9 (12.17) | -1.4 (12.90)
  Day 7 Observed: number analyzed (Participants) | 114 | 67 | 29 | 27 | 25 | 25 | 24 | 49 | 27
  Day 7 Observed | 72.9 (10.63) | 74.3 (9.90) | 71.5 (11.18) | 70.2 (10.40) | 70.0 (9.09) | 73.1 (9.62) | 69.8 (8.04) | 76.1 (9.30) | 71.8 (8.90)
  Day 7 Change: number analyzed (Participants) | 114 | 67 | 29 | 27 | 25 | 25 | 24 | 49 | 27
  Day 7 Change | -3.6 (11.56) | -3.5 (10.59) | -4.8 (12.01) | -6.9 (10.96) | -7.6 (10.25) | -4.5 (10.21) | -7.5 (12.94) | -2.6 (11.32) | -7.6 (14.12)
  Day 8 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 38
  Day 8 Observed |  |  |  |  |  |  |  | 73.5 (9.23) | 73.9 (11.18)
  Day 8 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 38
  Day 8 Change |  |  |  |  |  |  |  | -4.1 (10.98) | -3.5 (13.10)
  Day 9 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39 | 36
  Day 9 Observed |  |  |  |  |  |  |  | 75.5 (9.38) | 74.0 (11.92)
  Day 9 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39 | 36
  Day 9 Change |  |  |  |  |  |  |  | -1.7 (10.71) | -3.5 (12.63)
  Day 10 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 36 | 34
  Day 10 Observed |  |  |  |  |  |  |  | 74.6 (9.44) | 75.8 (12.46)
  Day 10 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 36 | 34
  Day 10 Change |  |  |  |  |  |  |  | -2.4 (9.31) | -1.2 (12.34)
  Day 11 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 28
  Day 11 Observed |  |  |  |  |  |  |  | 75.7 (10.37) | 76.3 (8.99)
  Day 11 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 28
  Day 11 Change |  |  |  |  |  |  |  | -0.9 (11.57) | -0.4 (10.87)
  Day 12 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 22
  Day 12 Observed |  |  |  |  |  |  |  | 77.3 (8.01) | 76.6 (8.26)
  Day 12 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 22
  Day 12 Change |  |  |  |  |  |  |  | 0.6 (10.39) | -0.5 (9.47)
  Day 13 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20
  Day 13 Observed |  |  |  |  |  |  |  | 77.2 (8.22) | 77.9 (8.98)
  Day 13 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20
  Day 13 Change |  |  |  |  |  |  |  | 1.3 (10.94) | 2.0 (13.71)
  Day 14 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0
  Day 14 Observed |  |  |  |  |  |  |  | 78.4 (7.81) |
  Day 14 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0
  Day 14 Change |  |  |  |  |  |  |  | 3.5 (9.72) |

9. Primary Outcome: Mean Observed and Change From Screening in Standing Diastolic Blood Pressure (mmHg): Vital Sign
Description: as for outcome 6
Time Frame: Day 1 to Day 14
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Inpatient: Pre 8AM | Inpatient: 3.5 hr Post 8AM | Inpatient: Pre 1PM | Inpatient: 3.5 hr Post 1PM | Inpatient: Pre 6PM | Inpatient: 3.5 hr Post 6PM | Inpatient: Pre 11PM | Outpatient: Predose | Outpatient: 3.5 hr Postdose
Number analyzed (Participants) | 286 | 286 | 286 | 286 | 286 | 286 | 286 | 286 | 286
mmHg
  Day 1 Observed: number analyzed (Participants) | 286 | 280 | 281 | 269 | 265 | 258 | 256 | 0 | 0
  Day 1 Observed | 79.8 (8.65) | 68.8 (11.34) | 70.3 (11.03) | 69.8 (11.87) | 70.7 (11.25) | 71.0 (11.12) | 70.4 (11.68) |  |
  Day 1 Change: number analyzed (Participants) | 0 | 279 | 281 | 268 | 264 | 257 | 255 | 0 | 0
  Day 1 Change |  | -11.1 (11.58) | -9.5 (11.26) | -10.0 (12.57) | -9.4 (11.73) | -8.9 (12.71) | -9.6 (12.92) |  |
  Day 2 Observed: number analyzed (Participants) | 251 | 235 | 226 | 218 | 216 | 212 | 213 | 0 | 0
  Day 2 Observed | 73.4 (11.02) | 70.7 (11.20) | 71.0 (11.48) | 71.6 (11.85) | 72.2 (11.78) | 72.3 (12.27) | 71.8 (11.52) |  |
  Day 2 Change: number analyzed (Participants) | 250 | 234 | 225 | 217 | 215 | 211 | 212 | 0 | 0
  Day 2 Change | -6.5 (11.83) | -9.4 (12.26) | -9.1 (12.74) | -8.5 (12.48) | -7.9 (13.00) | -7.9 (13.44) | -8.4 (13.05) |  |
  Day 3 Observed: number analyzed (Participants) | 213 | 207 | 206 | 203 | 203 | 203 | 201 | 0 | 0
  Day 3 Observed | 74.0 (12.03) | 70.6 (11.90) | 70.0 (10.53) | 70.0 (10.62) | 70.8 (10.77) | 71.3 (10.69) | 71.5 (10.90) |  |
  Day 3 Change: number analyzed (Participants) | 212 | 206 | 205 | 202 | 202 | 202 | 200 | 0 | 0
  Day 3 Change | -6.2 (12.37) | -9.4 (13.09) | -10.0 (11.74) | -10.1 (11.91) | -9.3 (12.00) | -8.8 (11.91) | -8.7 (11.78) |  |
  Day 4 Observed: number analyzed (Participants) | 161 | 158 | 149 | 144 | 140 | 137 | 133 | 39 | 37
  Day 4 Observed | 73.2 (11.80) | 70.6 (11.11) | 71.2 (11.12) | 71.5 (10.98) | 72.2 (10.59) | 71.2 (11.09) | 71.8 (10.14) | 75.7 (10.45) | 70.1 (10.26)
  Day 4 Change: number analyzed (Participants) | 160 | 157 | 148 | 143 | 139 | 136 | 132 | 39 | 37
  Day 4 Change | -7.0 (12.08) | -9.4 (11.90) | -9.2 (11.96) | -8.9 (12.91) | -8.0 (11.71) | -9.0 (12.64) | -8.2 (11.46) | -4.5 (13.21) | -10.0 (11.81)
  Day 5 Observed: number analyzed (Participants) | 134 | 134 | 132 | 132 | 131 | 129 | 129 | 50 | 46
  Day 5 Observed | 72.4 (10.04) | 70.0 (10.46) | 70.7 (10.76) | 70.3 (10.99) | 71.1 (11.38) | 70.2 (11.20) | 71.1 (10.94) | 74.8 (9.79) | 74.5 (10.44)
  Day 5 Change: number analyzed (Participants) | 133 | 133 | 131 | 131 | 130 | 128 | 128 | 50 | 46
  Day 5 Change | -7.6 (11.99) | -10.0 (11.47) | -9.2 (12.07) | -9.6 (13.00) | -8.7 (12.76) | -9.8 (12.01) | -9.0 (11.39) | -5.5 (10.70) | -6.3 (12.07)
  Day 6 Observed: number analyzed (Participants) | 127 | 126 | 122 | 122 | 121 | 120 | 119 | 50 | 44
  Day 6 Observed | 72.9 (10.11) | 69.3 (10.11) | 71.1 (10.70) | 70.2 (11.15) | 71.4 (11.43) | 72.1 (12.37) | 72.5 (11.07) | 74.1 (12.33) | 73.2 (11.31)
  Day 6 Change: number analyzed (Participants) | 126 | 125 | 121 | 121 | 120 | 119 | 118 | 50 | 44
  Day 6 Change | -7.1 (11.40) | -10.7 (12.20) | -8.9 (11.60) | -9.8 (12.77) | -8.6 (12.26) | -7.9 (13.33) | -7.5 (11.88) | -6.1 (13.61) | -6.8 (14.08)
  Day 7 Observed: number analyzed (Participants) | 114 | 67 | 29 | 27 | 25 | 25 | 24 | 49 | 27
  Day 7 Observed | 73.6 (11.16) | 73.2 (11.07) | 70.3 (11.17) | 71.3 (11.69) | 70.4 (11.25) | 72.5 (10.89) | 69.0 (8.93) | 77.1 (11.43) | 70.8 (11.27)
  Day 7 Change: number analyzed (Participants) | 113 | 66 | 28 | 26 | 24 | 24 | 23 | 49 | 27
  Day 7 Change | -6.2 (12.37) | -7.4 (11.17) | -9.5 (9.83) | -9.7 (12.29) | -10.8 (11.06) | -8.5 (12.94) | -11.8 (11.89) | -3.3 (12.24) | -10.4 (15.57)
  Day 8 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 38
  Day 8 Observed |  |  |  |  |  |  |  | 74.6 (9.22) | 74.5 (13.60)
  Day 8 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 38
  Day 8 Change |  |  |  |  |  |  |  | -5.8 (10.46) | -6.2 (14.23)
  Day 9 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39 | 36
  Day 9 Observed |  |  |  |  |  |  |  | 78.4 (9.63) | 76.5 (14.02)
  Day 9 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39 | 36
  Day 9 Change |  |  |  |  |  |  |  | -1.8 (10.89) | -4.2 (13.95)
  Day 10 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 36 | 34
  Day 10 Observed |  |  |  |  |  |  |  | 76.9 (10.41) | 75.9 (11.86)
  Day 10 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 36 | 34
  Day 10 Change |  |  |  |  |  |  |  | -3.2 (10.32) | -4.5 (12.68)
  Day 11 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 28
  Day 11 Observed |  |  |  |  |  |  |  | 78.1 (11.01) | 76.0 (9.55)
  Day 11 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 28
  Day 11 Change |  |  |  |  |  |  |  | -1.7 (10.96) | -3.9 (9.81)
  Day 12 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 22
  Day 12 Observed |  |  |  |  |  |  |  | 80.0 (8.12) | 78.7 (9.55)
  Day 12 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 22
  Day 12 Change |  |  |  |  |  |  |  | 0.3 (8.62) | -1.6 (11.95)
  Day 13 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20
  Day 13 Observed |  |  |  |  |  |  |  | 83.6 (8.38) | 80.8 (8.69)
  Day 13 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20
  Day 13 Change |  |  |  |  |  |  |  | 4.5 (10.29) | 1.1 (12.01)
  Day 14 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0
  Day 14 Observed |  |  |  |  |  |  |  | 84.8 (8.53) |
  Day 14 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0
  Day 14 Change |  |  |  |  |  |  |  | 5.5 (9.72) |

10. Primary Outcome: Mean Observed and Change From Screening in Seated Pulse (Bpm): Vital Signs
Description: as for outcome 6
Time Frame: Day 1 to Day 14
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Inpatient: Pre 8AM | Inpatient: 3.5 hr Post 8AM | Inpatient: Pre 1PM | Inpatient: 3.5 hr Post 1PM | Inpatient: Pre 6PM | Inpatient: 3.5 hr Post 6PM | Inpatient: Pre 11PM | Outpatient: Predose | Outpatient: 3.5 hr Postdose
Number analyzed (Participants) | 286 | 286 | 286 | 286 | 286 | 286 | 286 | 286 | 286
beats per minute (bpm)
  Day 1 Observed: number analyzed (Participants) | 286 | 285 | 283 | 270 | 266 | 259 | 256 | 0 | 0
  Day 1 Observed | 73.3 (10.89) | 68.8 (11.92) | 69.2 (11.08) | 69.9 (12.57) | 70.5 (12.28) | 67.6 (12.55) | 67.7 (12.08) |  |
  Day 1 Change: number analyzed (Participants) | 286 | 285 | 283 | 270 | 266 | 259 | 256 | 0 | 0
  Day 1 Change | NA (NA) — Prior to first dose. | -6.1 (12.75) | -5.7 (12.11) | -4.9 (13.47) | -4.3 (13.63) | -7.3 (13.59) | -7.0 (12.82) |  |
  Day 2 Observed: number analyzed (Participants) | 251 | 234 | 226 | 218 | 217 | 214 | 213 | 0 | 0
  Day 2 Observed | 70.2 (12.70) | 68.8 (12.36) | 69.4 (11.57) | 66.8 (12.65) | 68.7 (12.11) | 65.9 (12.41) | 66.4 (12.55) |  |
  Day 2 Change: number analyzed (Participants) | 251 | 234 | 226 | 218 | 217 | 214 | 213 | 0 | 0
  Day 2 Change | -4.7 (14.21) | -5.9 (14.63) | -5.4 (13.64) | -8.0 (14.53) | -6.2 (13.75) | -9.1 (14.30) | -8.6 (14.30) |  |
  Day 3 Observed: number analyzed (Participants) | 213 | 208 | 206 | 203 | 203 | 203 | 202 | 0 | 0
  Day 3 Observed | 213 (70.0) | 67.5 (12.97) | 68.7 (11.57) | 66.6 (12.03) | 68.3 (12.23) | 65.9 (11.68) | 67.4 (12.01) |  |
  Day 3 Change: number analyzed (Participants) | 213 | 208 | 206 | 203 | 203 | 203 | 202 | 0 | 0
  Day 3 Change | -5.0 (15.10) | -7.5 (15.52) | -6.4 (14.42) | -8.5 (14.77) | -6.8 (14.26) | -9.2 (14.25) | -7.8 (13.70) |  |
  Day 4 Observed: number analyzed (Participants) | 161 | 158 | 149 | 144 | 140 | 137 | 133 | 39 | 37
  Day 4 Observed | 70.1 (13.60) | 68.3 (12.46) | 70.6 (12.98) | 67.8 (13.00) | 70.0 (12.01) | 67.8 (13.80) | 69.9 (12.80) | 70.6 (11.83) | 72.4 (12.46)
  Day 4 Change: number analyzed (Participants) | 161 | 158 | 149 | 144 | 140 | 137 | 133 | 39 | 37
  Day 4 Change | -5.0 (16.11) | -6.8 (15.56) | -4.5 (15.43) | -7.3 (15.44) | -5.0 (15.35) | -6.8 (16.59) | -4.5 (14.74) | -5.2 (13.76) | -3.3 (13.25)
  Day 5 Observed: number analyzed (Participants) | 134 | 134 | 132 | 132 | 131 | 129 | 129 | 50 | 46
  Day 5 Observed | 70.9 (13.70) | 69.1 (11.03) | 71.4 (11.78) | 69.0 (13.35) | 68.7 (11.08) | 68.3 (12.84) | 70.0 (11.20) | 76.3 (13.49) | 73.3 (11.44)
  Day 5 Change: number analyzed (Participants) | 134 | 134 | 132 | 132 | 131 | 129 | 129 | 50 | 46
  Day 5 Change | -3.4 (16.28) | -5.3 (13.57) | -2.8 (13.92) | -5.2 (15.23) | -5.5 (12.29) | -6.0 (15.26) | -4.4 (13.53) | -0.3 (15.14) | -3.2 (13.70)
  Day 6 Observed: number analyzed (Participants) | 127 | 126 | 122 | 122 | 121 | 120 | 119 | 50 | 44
  Day 6 Observed | 70.5 (11.24) | 69.8 (12.46) | 70.6 (12.24) | 68.6 (11.43) | 69.7 (10.67) | 68.9 (13.05) | 71.2 (12.43) | 75.2 (12.24) | 74.8 (13.10)
  Day 6 Change: number analyzed (Participants) | 127 | 126 | 122 | 122 | 121 | 120 | 119 | 50 | 44
  Day 6 Change | -3.6 (14.98) | -4.1 (14.44) | -3.3 (13.62) | -5.3 (14.37) | -4.3 (12.88) | -5.1 (14.79) | -2.8 (13.55) | -1.6 (14.82) | -1.6 (14.29)
  Day 7 Observed: number analyzed (Participants) | 113 | 67 | 29 | 27 | 25 | 25 | 24 | 49 | 27
  Day 7 Observed | 73.2 (13.34) | 73.9 (11.70) | 73.6 (11.55) | 73.0 (12.53) | 73.6 (11.74) | 67.4 (13.44) | 69.8 (11.59) | 73.6 (11.46) | 67.1 (8.84)
  Day 7 Change: number analyzed (Participants) | 113 | 67 | 29 | 27 | 25 | 25 | 24 | 49 | 27
  Day 7 Change | -1.1 (16.86) | 0.0 (13.60) | -3.1 (13.15) | -3.8 (12.93) | -3.4 (11.72) | -9.5 (13.96) | 24 (13.29) | -3.4 (15.07) | -7.7 (10.63)
  Day 8 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 38
  Day 8 Observed |  |  |  |  |  |  |  | 77.7 (12.71) | 72.6 (13.45)
  Day 8 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 38
  Day 8 Change |  |  |  |  |  |  |  | 1.6 (15.25) | -3.8 (13.48)
  Day 9 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39 | 36
  Day 9 Observed |  |  |  |  |  |  |  | 79.6 (10.77) | 75.1 (11.19)
  Day 9 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39 | 36
  Day 9 Change |  |  |  |  |  |  |  | 2.8 (11.80) | -1.7 (11.18)
  Day 10 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 36 | 34
  Day 10 Observed |  |  |  |  |  |  |  | 80.0 (13.29) | 77.9 (16.42)
  Day 10 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 36 | 34
  Day 10 Change |  |  |  |  |  |  |  | 3.2 (14.82) | 1.1 (16.97)
  Day 11 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 28
  Day 11 Observed |  |  |  |  |  |  |  | 79.3 (13.93) | 74.5 (12.49)
  Day 11 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 28
  Day 11 Change |  |  |  |  |  |  |  | 3.2 (13.40) | -1.4 (12.92)
  Day 12 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 22
  Day 12 Observed |  |  |  |  |  |  |  | 79.7 (11.89) | 72.3 (11.68)
  Day 12 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 22
  Day 12 Change |  |  |  |  |  |  |  | 4.0 (14.22) | -3.6 (12.29)
  Day 13 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20
  Day 13 Observed |  |  |  |  |  |  |  | 76.6 (13.20) | 75.5 (13.61)
  Day 13 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20
  Day 13 Change |  |  |  |  |  |  |  | 2.4 (14.79) | 0.8 (11.75)
  Day 14 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0
  Day 14 Observed |  |  |  |  |  |  |  | 76.4 (11.66) |
  Day 14 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0
  Day 14 Change |  |  |  |  |  |  |  | 2.4 (14.27) |

11. Primary Outcome: Mean Observed and Change From Screening in Standing Pulse (Bpm): Vital Signs
Description: as for outcome 6
Time Frame: Day 1 to Day 14
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Inpatient: Pre 8AM | Inpatient: 3.5 hr Post 8AM | Inpatient: Pre 1PM | Inpatient: 3.5 hr Post 1PM | Inpatient: Pre 6PM | Inpatient: 3.5 hr Post 6PM | Inpatient: Pre 11PM | Outpatient: Predose | Outpatient: 3.5 hr Postdose
Number analyzed (Participants) | 286 | 286 | 286 | 286 | 286 | 286 | 286 | 286 | 286
beats per minute (bpm)
  Day 1 Observed: number analyzed (Participants) | 286 | 279 | 282 | 269 | 265 | 258 | 256 | 0 | 0
  Day 1 Observed | 82.8 (13.74) | 79.6 (14.29) | 80.1 (13.72) | 81.3 (14.42) | 81.2 (14.17) | 78.9 (14.14) | 79.4 (14.03) |  |
  Day 1 Change: number analyzed (Participants) | 286 | 279 | 282 | 269 | 265 | 258 | 256 | 0 | 0
  Day 1 Change | NA (NA) — Prior to first dose. | -1.8 (15.18) | -1.3 (14.38) | 0.0 (16.41) | -0.1 (15.89) | -2.5 (16.25) | -1.8 (16.00) |  |
  Day 2 Observed: number analyzed (Participants) | 251 | 234 | 226 | 218 | 217 | 212 | 213 | 0 | 0
  Day 2 Observed | 82.4 (15.13) | 80.6 (15.19) | 81.1 (13.74) | 80.5 (14.44) | 80.8 (14.46) | 78.0 (14.67) | 78.4 (13.95) |  |
  Day 2 Change: number analyzed (Participants) | 251 | 234 | 226 | 218 | 217 | 212 | 213 | 0 | 0
  Day 2 Change | 1.0 (16.81) | -0.5 (17.61) | 0.0 (16.22) | -0.6 (15.44) | -0.4 (16.00) | -3.3 (16.49) | -3.0 (16.62) |  |
  Day 3 Observed: number analyzed (Participants) | 213 | 207 | 206 | 203 | 203 | 203 | 200 | 0 | 0
  Day 3 Observed | 81.1 (14.82) | 79.0 (14.24) | 80.0 (14.67) | 78.1 (15.09) | 79.1 (15.36) | 76.4 (13.75) | 78.3 (13.92) |  |
  Day 3 Change: number analyzed (Participants) | 213 | 207 | 206 | 203 | 203 | 203 | 200 | 0 | 0
  Day 3 Change | -0.2 (16.77) | -2.6 (16.59) | -1.5 (15.95) | -3.3 (17.08) | -2.3 (16.27) | -5.0 (16.31) | -3.2 (16.32) |  |
  Day 4 Observed: number analyzed (Participants) | 161 | 158 | 149 | 144 | 140 | 137 | 132 | 39 | 37
  Day 4 Observed | 81.2 (14.93) | 80.1 (14.67) | 81.5 (15.40) | 79.9 (15.42) | 80.8 (16.34) | 78.2 (15.52) | 80.4 (16.16) | 82.0 (11.75) | 83.3 (15.43)
  Day 4 Change: number analyzed (Participants) | 161 | 158 | 149 | 144 | 140 | 137 | 132 | 39 | 37
  Day 4 Change | -0.2 (16.09) | -1.3 (16.36) | 0.0 (16.85) | -1.5 (17.75) | -0.7 (18.62) | -2.7 (17.29) | -0.2 (17.49) | 0.9 (15.06) | 2.1 (18.73)
  Day 5 Observed: number analyzed (Participants) | 134 | 134 | 132 | 132 | 131 | 129 | 129 | 50 | 46
  Day 5 Observed | 83.1 (16.31) | 81.0 (14.06) | 82.3 (15.43) | 84.7 (51.39) | 80.2 (14.86) | 79.5 (14.08) | 80.6 (14.74) | 85.2 (15.23) | 80.8 (14.81)
  Day 5 Change: number analyzed (Participants) | 134 | 134 | 132 | 132 | 131 | 129 | 129 | 50 | 46
  Day 5 Change | 2.4 (18.58) | 0.3 (15.33) | 1.6 (16.77) | 4.2 (50.96) | -0.4 (14.80) | -1.2 (15.68) | -0.1 (16.33) | 2.8 (16.75) | -1.7 (15.90)
  Day 6 Observed: number analyzed (Participants) | 127 | 126 | 122 | 122 | 121 | 120 | 119 | 50 | 44
  Day 6 Observed | 81.7 (14.96) | 79.9 (14.89) | 81.8 (14.90) | 79.5 (14.00) | 81.5 (13.93) | 80.9 (14.54) | 80.9 (15.77) | 86.4 (15.08) | 84.8 (14.77)
  Day 6 Change: number analyzed (Participants) | 127 | 126 | 122 | 122 | 121 | 120 | 119 | 50 | 44
  Day 6 Change | 1.4 (16.05) | -0.5 (16.33) | 1.4 (15.99) | -0.9 (16.16) | 1.0 (15.28) | 0.4 (15.68) | 0.4 (16.97) | 2.6 (16.42) | 1.6 (15.33)
  Day 7 Observed: number analyzed (Participants) | 113 | 67 | 29 | 27 | 25 | 25 | 24 | 49 | 27
  Day 7 Observed | 84.5 (15.44) | 80.3 (12.44) | 83.4 (13.89) | 79.0 (13.45) | 80.0 (14.40) | 75.1 (13.69) | 74.3 (12.41) | 83.2 (13.11) | 76.9 (11.29)
  Day 7 Change: number analyzed (Participants) | 113 | 67 | 29 | 27 | 25 | 25 | 24 | 49 | 27
  Day 7 Change | 3.5 (18.07) | 0.2 (14.16) | -0.5 (16.23) | -4.9 (14.53) | -3.6 (16.19) | -8.6 (17.80) | -9.7 (16.75) | -0.5 (16.99) | -4.3 (12.54)
  Day 8 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 38
  Day 8 Observed |  |  |  |  |  |  |  | 85.3 (15.03) | 80.7 (14.61)
  Day 8 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 38
  Day 8 Change |  |  |  |  |  |  |  | 2.5 (18.08) | -2.9 (15.07)
  Day 9 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39 | 36
  Day 9 Observed |  |  |  |  |  |  |  | 90.7 (16.51) | 82.8 (15.66)
  Day 9 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39 | 36
  Day 9 Change |  |  |  |  |  |  |  | 6.8 (15.74) | -1.1 (14.94)
  Day 10 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 36 | 34
  Day 10 Observed |  |  |  |  |  |  |  | 88.7 (15.73) | 85.1 (17.87)
  Day 10 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 36 | 34
  Day 10 Change |  |  |  |  |  |  |  | 5.1 (17.47) | 1.6 (18.66)
  Day 11 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 28
  Day 11 Observed |  |  |  |  |  |  |  | 89.3 (16.55) | 82.0 (16.84)
  Day 11 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 28
  Day 11 Change |  |  |  |  |  |  |  | 6.4 (16.75) | -0.1 (17.81)
  Day 12 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 22
  Day 12 Observed |  |  |  |  |  |  |  | 90.8 (16.25) | 80.0 (13.91)
  0Day 12 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 22
  0Day 12 Change |  |  |  |  |  |  |  | 9.2 (17.91) | -1.4 (16.75)
  Day 13 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20
  Day 13 Observed |  |  |  |  |  |  |  | 86.6 (13.51) | 81.4 (13.21)
  Day 13 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20
  Day 13 Change |  |  |  |  |  |  |  | 6.2 (17.17) | 1.1 (15.14)
  Day 14 Observed: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0
  Day 14 Observed |  |  |  |  |  |  |  | 87.0 (17.66) |
  Day 14 Change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 0
  Day 14 Change |  |  |  |  |  |  |  | 7.2 (19.63) |

12. Primary Outcome: Columbia Suicide Severity Rating Scale Questionnaire (C-SSRS): Suicidal Ideation and Behavior Numbers
Description: The C-SSRS measures both suicidal ideation and suicidal behavior and will be completed to assess lifetime suicidality before first dose of study drug, 3.5 hours after first daily dose of study drug on in-clinic treatment days, and then once a day before dosing during outpatient treatment days. C-SSRS will also be assessed at end of study/discontinuation.
Time Frame: Day 1 to Day 14
Population: Suicidality: The number and percentage of subjects reporting any suicidal ideation OR behavior throughout the assessment period, including baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | OL: Lofexidine HCl
Number analyzed (Participants) | 286
Participants
  Suicidality | 30
  Suicidal ideation | 27
  Suicidal behavior | 12
  Emergence of suicidal ideation | 2
  Emergence of serious suicidal ideation | 0
  Worsening of suicidal ideation | 2
  Emergence of suicidal behavior | 0

13. Primary Outcome: Clinical Laboratory Test Change From Baseline: Hematology
Description: Hematology Parameters with Shifts in ≥3% of Subjects from Screening to End of Study
Time Frame: Day 1 to Day 14
Population: The number of participants analyzed for each parameter differs from the overall number of participants analyzed as a result of missing data for some participants.
Measure: Count of Participants; unit: Participants
Groups:
- Below Baseline (End of Study): Shifts from normal at baseline to below baseline at the last post-baseline assessment for hematology parameters occurring in ≥3% of subjects.
  Lofexidine: All enrolled subjects will take lofexidine orally, starting on Day 1 at a dose of 3.2 mg per day (0.8 mg QID), with lowering of the dose allowed to 2.4 mg daily (0.6 mg QID) if required for tolerability based on the subject's individual treatment goal and response per clinical judgment of the Principal Investigator.
- Normal (End of Study): Subjects whose normal baseline hematology parameters did not shift below or above baseline at the last post-baseline assessment occurring in ≥3% of subjects.
  Lofexidine: All enrolled subjects will take lofexidine orally, starting on Day 1 at a dose of 3.2 mg per day (0.8 mg QID), with lowering of the dose allowed to 2.4 mg daily (0.6 mg QID) if required for tolerability based on the subject's individual treatment goal and response per clinical judgment of the Principal Investigator.
- Above Baseline (End of Study): Shifts from normal at baseline to above baseline at the last post-baseline assessment for hematology parameters occurring in ≥3% of subjects.
  Lofexidine: All enrolled subjects will take lofexidine orally, starting on Day 1 at a dose of 3.2 mg per day (0.8 mg QID), with lowering of the dose allowed to 2.4 mg daily (0.6 mg QID) if required for tolerability based on the subject's individual treatment goal and response per clinical judgment of the Principal Investigator.
Arm/Group | Below Baseline (End of Study) | Normal (End of Study) | Above Baseline (End of Study)
Number analyzed (Participants) | 286 | 286 | 286
Participants
  Hemoglobin (g/dL) : Below (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Hemoglobin (g/dL) : Below (Baseline) | 25 | 27 | 0
  Hemoglobin (g/dL) : Normal (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Hemoglobin (g/dL) : Normal (Baseline) | 8 | 124 | 8
  Hemoglobin (g/dL) : Above (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Hemoglobin (g/dL) : Above (Baseline) | 0 | 1 | 9
  Hematocrit (%) : Below (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Hematocrit (%) : Below (Baseline) | 11 | 23 | 0
  Hematocrit (%) : Normal (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Hematocrit (%) : Normal (Baseline) | 6 | 120 | 20
  Hematocrit (%) : Above (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Hematocrit (%) : Above (Baseline) | 0 | 10 | 12
  Platelet count (x10^9/L) : Below (Baseline): number analyzed (Participants) | 197 | 197 | 197
  Platelet count (x10^9/L) : Below (Baseline) | 11 | 0 | 0
  Platelet count (x10^9/L) : Normal (Baseline): number analyzed (Participants) | 197 | 197 | 197
  Platelet count (x10^9/L) : Normal (Baseline) | 4 | 166 | 10
  Platelet count (x10^9/L) : Above (Baseline): number analyzed (Participants) | 197 | 197 | 197
  Platelet count (x10^9/L) : Above (Baseline) | 0 | 4 | 2
  Erythrocytes (x10^12/L) : Below (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Erythrocytes (x10^12/L) : Below (Baseline) | 14 | 20 | 0
  Erythrocytes (x10^12/L) : Normal (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Erythrocytes (x10^12/L) : Normal (Baseline) | 11 | 122 | 16
  Erythrocytes (x10^12/L) : Above (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Erythrocytes (x10^12/L) : Above (Baseline) | 0 | 8 | 11
  Erythrocytes distribution width (%) : Below (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Erythrocytes distribution width (%) : Below (Baseline) | 0 | 0 | 0
  Erythrocytes distribution width (%) : Normal (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Erythrocytes distribution width (%) : Normal (Baseline) | 0 | 150 | 22
  Erythrocytes distribution width (%) : Above (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Erythrocytes distribution width (%) : Above (Baseline) | 0 | 8 | 22
  Mean corpuscular volume (fL) : Below (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Mean corpuscular volume (fL) : Below (Baseline) | 4 | 2 | 0
  Mean corpuscular volume (fL) : Normal (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Mean corpuscular volume (fL) : Normal (Baseline) | 0 | 173 | 6
  Mean corpuscular volume (fL) : Above (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Mean corpuscular volume (fL) : Above (Baseline) | 0 | 4 | 13
  Leukocytes (x10^9/L) : Below (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Leukocytes (x10^9/L) : Below (Baseline) | 0 | 2 | 0
  Leukocytes (x10^9/L) : Normal (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Leukocytes (x10^9/L) : Normal (Baseline) | 2 | 167 | 23
  Leukocytes (x10^9/L) : Above (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Leukocytes (x10^9/L) : Above (Baseline) | 0 | 4 | 4
  Neutrophils/Leukocytes (%) : Below (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Neutrophils/Leukocytes (%) : Below (Baseline) | 0 | 4 | 0
  Neutrophils/Leukocytes (%) : Normal (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Neutrophils/Leukocytes (%) : Normal (Baseline) | 2 | 163 | 19
  Neutrophils/Leukocytes (%) : Above (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Neutrophils/Leukocytes (%) : Above (Baseline) | 0 | 8 | 6
  Neutrophils (x10^9/L) : Below (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Neutrophils (x10^9/L) : Below (Baseline) | 0 | 0 | 0
  Neutrophils (x10^9/L) : Normal (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Neutrophils (x10^9/L) : Normal (Baseline) | 1 | 182 | 13
  Neutrophils (x10^9/L) : Above (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Neutrophils (x10^9/L) : Above (Baseline) | 0 | 3 | 3
  Lymphocytes/Leukocytes (%) : Below (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Lymphocytes/Leukocytes (%) : Below (Baseline) | 23 | 15 | 1
  Lymphocytes/Leukocytes (%) : Normal (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Lymphocytes/Leukocytes (%) : Normal (Baseline) | 32 | 103 | 10
  Lymphocytes/Leukocytes (%) : Above (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Lymphocytes/Leukocytes (%) : Above (Baseline) | 1 | 12 | 5
  Lymphocytes, absolute (x10^9/L) : Below (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Lymphocytes, absolute (x10^9/L) : Below (Baseline) | 1 | 2 | 0
  Lymphocytes, absolute (x10^9/L) : Normal (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Lymphocytes, absolute (x10^9/L) : Normal (Baseline) | 3 | 192 | 2
  Lymphocytes, absolute (x10^9/L) : Above (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Lymphocytes, absolute (x10^9/L) : Above (Baseline) | 0 | 1 | 1
  Monocytes/Leukocytes (%) : Below (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Monocytes/Leukocytes (%) : Below (Baseline) | 0 | 0 | 0
  Monocytes/Leukocytes (%) : Normal (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Monocytes/Leukocytes (%) : Normal (Baseline) | 1 | 159 | 19
  Monocytes/Leukocytes (%) : Above (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Monocytes/Leukocytes (%) : Above (Baseline) | 0 | 17 | 6
  Monocytes (x10^9/L) : Below (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Monocytes (x10^9/L) : Below (Baseline) | 0 | 0 | 0
  Monocytes (x10^9/L) : Normal (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Monocytes (x10^9/L) : Normal (Baseline) | 0 | 192 | 7
  Monocytes (x10^9/L) : Above (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Monocytes (x10^9/L) : Above (Baseline) | 0 | 2 | 1
  Eosinophils absolute (x10^9/L) : Below (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Eosinophils absolute (x10^9/L) : Below (Baseline) | 0 | 0 | 0
  Eosinophils absolute (x10^9/L) : Normal (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Eosinophils absolute (x10^9/L) : Normal (Baseline) | 0 | 176 | 9
  Eosinophils absolute (x10^9/L) : Above (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Eosinophils absolute (x10^9/L) : Above (Baseline) | 0 | 10 | 7
  Eosinophils/Leukocytes (%) : Below (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Eosinophils/Leukocytes (%) : Below (Baseline) | 0 | 0 | 0
  Eosinophils/Leukocytes (%) : Normal (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Eosinophils/Leukocytes (%) : Normal (Baseline) | 0 | 140 | 12
  Eosinophils/Leukocytes (%) : Above (Baseline): number analyzed (Participants) | 202 | 202 | 202
  Eosinophils/Leukocytes (%) : Above (Baseline) | 0 | 31 | 19
  Prothrombin time (seconds) : Below (Baseline): number analyzed (Participants) | 205 | 205 | 205
  Prothrombin time (seconds) : Below (Baseline) | 0 | 0 | 0
  Prothrombin time (seconds) : Normal (Baseline): number analyzed (Participants) | 205 | 205 | 205
  Prothrombin time (seconds) : Normal (Baseline) | 0 | 154 | 20
  Prothrombin time (seconds) : Above (Baseline): number analyzed (Participants) | 205 | 205 | 205
  Prothrombin time (seconds) : Above (Baseline) | 0 | 17 | 14
  Activated Partial Thromboplastin Time (seconds) : Below (Baseline): number analyzed (Participants) | 205 | 205 | 205
  Activated Partial Thromboplastin Time (seconds) : Below (Baseline) | 0 | 1 | 0
  Activated Partial Thromboplastin Time (seconds) : Normal (Baseline): number analyzed (Participants) | 205 | 205 | 205
  Activated Partial Thromboplastin Time (seconds) : Normal (Baseline) | 0 | 154 | 13
  Activated Partial Thromboplastin Time (seconds) : Above (Baseline): number analyzed (Participants) | 205 | 205 | 205
  Activated Partial Thromboplastin Time (seconds) : Above (Baseline) | 0 | 19 | 18

14. Primary Outcome: Clinical Laboratory Test Change From Baseline: Chemistry
Description: Chemistry Parameters with Shifts in ≥3% of Subjects from Screening to End of Study
Time Frame: Day 1 to Day 14
Population: Participants Analyzed does not match the Participant Flow as a result of missing data for some participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Below Baseline (End of Study) | Normal (End of Study) | Above Baseline (End of Study)
Number analyzed (Participants) | 286 | 286 | 286
Participants
  Alanine aminotransferase (U/L) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Alanine aminotransferase (U/L) : Below (Baseline) | 0 | 0 | 0
  Alanine aminotransferase (U/L) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Alanine aminotransferase (U/L) : Normal (Baseline) | 0 | 153 | 17
  Alanine aminotransferase (U/L) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Alanine aminotransferase (U/L) : Above (Baseline) | 0 | 12 | 22
  Aspartate Aminotransferase (U/L) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Aspartate Aminotransferase (U/L) : Below (Baseline) | 0 | 0 | 0
  Aspartate Aminotransferase (U/L) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Aspartate Aminotransferase (U/L) : Normal (Baseline) | 0 | 164 | 10
  Aspartate Aminotransferase (U/L) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Aspartate Aminotransferase (U/L) : Above (Baseline) | 0 | 16 | 14
  Gamma-glutamyl transferase (U/L) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Gamma-glutamyl transferase (U/L) : Below (Baseline) | 9 | 13 | 0
  Gamma-glutamyl transferase (U/L) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Gamma-glutamyl transferase (U/L) : Normal (Baseline) | 2 | 139 | 11
  Gamma-glutamyl transferase (U/L) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Gamma-glutamyl transferase (U/L) : Above (Baseline) | 0 | 6 | 24
  Alkaline phosphatase (U/L) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Alkaline phosphatase (U/L) : Below (Baseline) | 6 | 3 | 0
  Alkaline phosphatase (U/L) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Alkaline phosphatase (U/L) : Normal (Baseline) | 9 | 170 | 3
  Alkaline phosphatase (U/L) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Alkaline phosphatase (U/L) : Above (Baseline) | 0 | 5 | 8
  Lactate dehydrogenase (U/L) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Lactate dehydrogenase (U/L) : Below (Baseline) | 2 | 0 | 0
  Lactate dehydrogenase (U/L) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Lactate dehydrogenase (U/L) : Normal (Baseline) | 3 | 164 | 7
  Lactate dehydrogenase (U/L) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Lactate dehydrogenase (U/L) : Above (Baseline) | 0 | 19 | 9
  Blood urea nitrogen (mg/dL) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Blood urea nitrogen (mg/dL) : Below (Baseline) | 9 | 28 | 1
  Blood urea nitrogen (mg/dL) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Blood urea nitrogen (mg/dL) : Normal (Baseline) | 28 | 127 | 5
  Blood urea nitrogen (mg/dL) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Blood urea nitrogen (mg/dL) : Above (Baseline) | 1 | 4 | 1
  Creatinine (mg/dL) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Creatinine (mg/dL) : Below (Baseline) | 29 | 17 | 0
  Creatinine (mg/dL) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Creatinine (mg/dL) : Normal (Baseline) | 8 | 147 | 2
  Creatinine (mg/dL) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Creatinine (mg/dL) : Above (Baseline) | 0 | 0 | 1
  Cholesterol (mg/dL) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Cholesterol (mg/dL) : Below (Baseline) | 0 | 0 | 0
  Cholesterol (mg/dL) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Cholesterol (mg/dL) : Normal (Baseline) | 0 | 153 | 18
  Cholesterol (mg/dL) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Cholesterol (mg/dL) : Above (Baseline) | 0 | 13 | 20
  Triglycerides (mg/dL) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Triglycerides (mg/dL) : Below (Baseline) | 0 | 0 | 0
  Triglycerides (mg/dL) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Triglycerides (mg/dL) : Normal (Baseline) | 0 | 107 | 40
  Triglycerides (mg/dL) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Triglycerides (mg/dL) : Above (Baseline) | 0 | 18 | 39
  Calcium (mg/dL) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Calcium (mg/dL) : Below (Baseline) | 1 | 9 | 0
  Calcium (mg/dL) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Calcium (mg/dL) : Normal (Baseline) | 7 | 182 | 3
  Calcium (mg/dL) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Calcium (mg/dL) : Above (Baseline) | 0 | 2 | 0
  Sodium (mEq/L) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Sodium (mEq/L) : Below (Baseline) | 3 | 6 | 0
  Sodium (mEq/L) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Sodium (mEq/L) : Normal (Baseline) | 3 | 187 | 5
  Sodium (mEq/L) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Sodium (mEq/L) : Above (Baseline) | 0 | 0 | 0
  Potassium (mEq/L) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Potassium (mEq/L) : Below (Baseline) | 0 | 2 | 0
  Potassium (mEq/L) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Potassium (mEq/L) : Normal (Baseline) | 2 | 183 | 11
  Potassium (mEq/L) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Potassium (mEq/L) : Above (Baseline) | 0 | 6 | 0
  Chloride (mEq/L) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Chloride (mEq/L) : Below (Baseline) | 0 | 5 | 0
  Chloride (mEq/L) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Chloride (mEq/L) : Normal (Baseline) | 3 | 190 | 5
  Chloride (mEq/L) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Chloride (mEq/L) : Above (Baseline) | 0 | 0 | 1
  Carbon dioxide (bicarbonate) (mEq/L) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Carbon dioxide (bicarbonate) (mEq/L) : Below (Baseline) | 0 | 0 | 0
  Carbon dioxide (bicarbonate) (mEq/L) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Carbon dioxide (bicarbonate) (mEq/L) : Normal (Baseline) | 3 | 134 | 7
  Carbon dioxide (bicarbonate) (mEq/L) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Carbon dioxide (bicarbonate) (mEq/L) : Above (Baseline) | 0 | 52 | 8
  Glucose (mg/dL) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Glucose (mg/dL) : Below (Baseline) | 0 | 5 | 0
  Glucose (mg/dL) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Glucose (mg/dL) : Normal (Baseline) | 1 | 130 | 35
  Glucose (mg/dL) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Glucose (mg/dL) : Above (Baseline) | 0 | 19 | 14
  Phosphate (mg/dL) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Phosphate (mg/dL) : Below (Baseline) | 1 | 4 | 0
  Phosphate (mg/dL) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Phosphate (mg/dL) : Normal (Baseline) | 6 | 138 | 22
  Phosphate (mg/dL) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Phosphate (mg/dL) : Above (Baseline) | 1 | 26 | 6
  Protein (g/dL) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Protein (g/dL) : Below (Baseline) | 0 | 1 | 0
  Protein (g/dL) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Protein (g/dL) : Normal (Baseline) | 0 | 190 | 4
  Protein (g/dL) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Protein (g/dL) : Above (Baseline) | 0 | 6 | 3
  Thyroid Stimulating Hormone-3rd Generation (TSH Thyrotropin)(mU/L) : Below (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Thyroid Stimulating Hormone-3rd Generation (TSH Thyrotropin)(mU/L) : Below (Baseline) | 11 | 18 | 0
  Thyroid Stimulating Hormone-3rd Generation (TSH Thyrotropin)(mU/L) : Normal (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Thyroid Stimulating Hormone-3rd Generation (TSH Thyrotropin)(mU/L) : Normal (Baseline) | 16 | 149 | 3
  Thyroid Stimulating Hormone-3rd Generation (TSH Thyrotropin)(mU/L) : Above (Baseline): number analyzed (Participants) | 204 | 204 | 204
  Thyroid Stimulating Hormone-3rd Generation (TSH Thyrotropin)(mU/L) : Above (Baseline) | 0 | 6 | 1

15. Primary Outcome: Clinical Laboratory Test Change From Baseline: Urinalysis
Time Frame: Day 1 to Day 7
Population: Participants Analyzed does not match the Participant Flow as a result of missing data for some participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Below Baseline (End of Study) | Normal (End of Study) | Above Baseline (End of Study)
Number analyzed (Participants) | 286 | 286 | 286
Participants
  Erythrocytes (/HPF) : Below (Baseline): number analyzed (Participants) | 207 | 207 | 207
  Erythrocytes (/HPF) : Below (Baseline) | 0 | 0 | 0
  Erythrocytes (/HPF) : Normal (Baseline): number analyzed (Participants) | 207 | 207 | 207
  Erythrocytes (/HPF) : Normal (Baseline) | 0 | 136 | 30
  Erythrocytes (/HPF) : Above (Baseline): number analyzed (Participants) | 207 | 207 | 207
  Erythrocytes (/HPF) : Above (Baseline) | 0 | 28 | 13
  Leukocytes (/HPF) : Below (Baseline): number analyzed (Participants) | 207 | 207 | 207
  Leukocytes (/HPF) : Below (Baseline) | 0 | 0 | 0
  Leukocytes (/HPF) : Normal (Baseline): number analyzed (Participants) | 207 | 207 | 207
  Leukocytes (/HPF) : Normal (Baseline) | 0 | 175 | 15
  Leukocytes (/HPF) : Above (Baseline): number analyzed (Participants) | 207 | 207 | 207
  Leukocytes (/HPF) : Above (Baseline) | 0 | 13 | 4
  Specific Gravity : Below (Baseline): number analyzed (Participants) | 207 | 207 | 207
  Specific Gravity : Below (Baseline) | 0 | 2 | 0
  Specific Gravity : Normal (Baseline): number analyzed (Participants) | 207 | 207 | 207
  Specific Gravity : Normal (Baseline) | 0 | 188 | 3
  Specific Gravity : Above (Baseline): number analyzed (Participants) | 207 | 207 | 207
  Specific Gravity : Above (Baseline) | 0 | 13 | 1
  pH : Below (Baseline): number analyzed (Participants) | 207 | 207 | 207
  pH : Below (Baseline) | 0 | 0 | 0
  pH : Normal (Baseline): number analyzed (Participants) | 207 | 207 | 207
  pH : Normal (Baseline) | 0 | 204 | 1
  pH : Above (Baseline): number analyzed (Participants) | 207 | 207 | 207
  pH : Above (Baseline) | 0 | 2 | 0

16. Primary Outcome: Safety Electrocardiograms (ECG) Evaluation Shift From Baseline to Post Dose and End of Study
Description: For each 12-lead ECG obtained during the study, the investigator made an overall interpretation of the ECG (normal, abnormal NCS, and abnormal CS). Shifts from normal at baseline to abnormal NCS and abnormal CS at the end of study predose and postdose assessments were summarized.
Time Frame: Day 1 and Day 14
Population: Participants Analyzed does not match the Participant Flow as a result of missing data for some participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Finding: Normal (OL: Lofexidine HCl) | Baseline Finding: Abnormal (NCS) (OL: Lofexidine HCl) | Baseline Finding: Abnormal (CS) (OL: Lofexidine HCl) | Total (OL: Lofexidine HCl)
Number analyzed (Participants) | 180 | 103 | 0 | 283
Participants
  Day 1 Post 8am Dose: Normal | 139 | 16 | 0 | 155
  Day 1 Post 8am Dose: Abnormal (NCS) | 41 | 87 | 0 | 128
  Day 1 Post 8am Dose: Abnormal (CS) | 0 | 0 | 0 | 0
  End of Study Pre Dose: number analyzed (Participants) | 103 | 58 | 0 | 161
  End of Study Pre Dose: Normal | 83 | 20 | 0 | 103
  End of Study Pre Dose: Abnormal (NCS) | 19 | 38 | 0 | 57
  End of Study Pre Dose: Abnormal (CS) | 1 | 0 | 0 | 1
  End of Study Post Dose: number analyzed (Participants) | 120 | 73 | 0 | 193
  End of Study Post Dose: Normal | 77 | 26 | 0 | 103
  End of Study Post Dose: Abnormal (NCS) | 41 | 47 | 0 | 88
  End of Study Post Dose: Abnormal (CS) | 2 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: AEs will be followed starting with dosing on Day 1 through Day 14, and will be evaluated as well on a 30-day post-last dose follow-up phone call.
Arm/Group | OL: Lofexidine HCl
All-Cause Mortality (participants affected / at risk) | 0/286
Serious Adverse Events (participants affected / at risk) | 2/286
Other Adverse Events (participants affected / at risk) | 270/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OL: Lofexidine HCl (N=286)
Delusion (Psychiatric disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OL: Lofexidine HCl (N=286)
Insomnia (Psychiatric disorders) | 144
Anxiety (Psychiatric disorders) | 107
Orthostatic hypotension (Vascular disorders) | 96
Hypotension (Vascular disorders) | 84
Bradycardia (Cardiac disorders) | 72
Diarrhea (Gastrointestinal disorders) | 54
Sedation (Nervous system disorders) | 46
Headache (Nervous system disorders) | 43
Abdominal pain upper (Gastrointestinal disorders) | 42
Myalgia (Musculoskeletal and connective tissue disorders) | 41
Constipation (Gastrointestinal disorders) | 15
Dry Mouth (Gastrointestinal disorders) | 24
Vomiting (Gastrointestinal disorders) | 26
Pain (General disorders) | 24
Somnolence (Nervous system disorders) | 21
Restlessness (Psychiatric disorders) | 22
Fatigue (General disorders) | 19
Back pain (Musculoskeletal and connective tissue disorders) | 15
Nausea (Gastrointestinal disorders) | 50
Dizziness (Nervous system disorders) | 47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2015-05-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT02363998/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT02363998/SAP_001.pdf
  • Informed Consent Form (2015-01-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT02363998/ICF_002.pdf